CLINICAL TRIAL: NCT05559697
Title: Healthy Human Study on DeRoyal Incisional Dressing With NPWT Compared Against Standard of Care NPWT Incision Dressing to Investigate Bioburden Levels and Skin Condition After Seven Day Period
Brief Title: Study Comparing iNPWT Dressing and Devices Affect on Bioburden Levels and Skin Condition After Seven Days
Acronym: HHiNPWT7DC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DeRoyal Industries, Inc. (Industry)
Collaborators: Lincoln Memorial University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1139
Record Dates: First submitted 2022-09-09; First posted 2022-09-29 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Skin Reaction to Mechanical, Thermal and Radiation Stimuli; Skin Sensitisation
Keywords: skin flora; incisional negative pressure wound therapy; dressing survivability
MeSH Terms: interventions — Bandages

STUDY DESIGN:
Intervention Model Description: Healthy human knees are prepped as if for total knee replacement. Incisional negative pressure dressings are applied to both knees.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Clinician research performing skin assessment masked from knee assignment to two interventions. Before the assessment, a separate clinician will remove the dressings and perform other measurements. The investigator performing data analysis will not know group assignment until unblinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Prospera Flex Incisional NPWT System (Experimental): Sponsor incisional dressing connected to sponsor disposable negative pressure device placed on knee for seven days.
  Interventions: Device: Sponsor incisional negative pressure wound therapy device and dressing
- Prevena Incisional NPWT System (Active Comparator): Market leader incisional NPWT system (includes the device and dressing) placed on opposite knee for seven days.
  Interventions: Device: Standard of Care incisional negative pressure wound therapy system

INTERVENTIONS:
Device: Sponsor incisional negative pressure wound therapy device and dressing — A sponsor incisional dressing placed on the knee and connected to a sponsor disposable negative pressure therapy device
  Arms: Prospera Flex Incisional NPWT System
Device: Standard of Care incisional negative pressure wound therapy system — The control incisional negative pressure wound therapy system represents the standard of care system and market leader. It consists of a disposable negative pressure therapy device and incisional dressing.
  Arms: Prevena Incisional NPWT System

SUMMARY:
Incisional dressings aim to prevent contamination of an incisional wound and protect against skin irritation. Surgeons use incisional negative pressure wound therapy (iNPWT) to manage incisional wounds. This study compares a new dressing designed for use with iNPWT that aims to improve comfort, tolerability, and dressing survivability over the standard of care for iNPWT. Further, no evidence exists that shows NPWT reduces the bacterial burden on the skin. This study will compare the incidence of skin irritation, dressing damage or lift, and changes in bacteria flora on healthy volunteer skin.

DETAILED DESCRIPTION:
The study compares the DeRoyal Negative Pressure Wound Therapy Incisional Dressing used with the DeRoyal Disposable NPWT device (experimental) to the market leader NPWT Incision Dressing system (control) over seven days to compare skin flora rebound, dressing degradation, skin irritation, and overall user experience. The protocol simulates the preparation of both knees for total knee replacement surgery (Day 0). After prepping the knee (shaving and chlorohexidine gluconate scrub), research personnel will swab the knee cap for an initial bioburden assessment. One knee is randomized to receive the experimental intervention, and the other knee receives the control intervention. Participants will wear both dressings for seven days documenting interruptions in the NPWT for activities of daily living, system-related discomfort, self-assessment of dressing damage, and tolerance for each system. Participants return to the clinic after seven days. First, research personnel will document each dressing's condition with photography and an assessment scale. The research staff will remove dressings under aseptic conditions, photograph each knee, and swab each for bioburden analysis. A blinded researcher will assess each knee for skin redness, irritation, blistering, or other skin adverse event and overall appearance using an adapted FDA scale for skin irritation. The participant's participation in the trial ends at this point. The resulting data will be analyzed using statistical methods to inform on differences in bioburden present under each dressing, the incidence of skin irritation or other adverse events, dressing survivability, discomfort differences, and tolerance of each system.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, aged 40 to 80 years of age
4. In good general health as evidenced by medical history
5. Healthy skin located across both knees at the dressing site location
6. No history of chronic knee pain
7. For females of reproductive potential: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study
8. Agreement to adhere to Lifestyle limitations throughout study duration
9. Ability to understand and write in English

Exclusion Criteria:

1. The presence of localized skin conditions, such as scaring, local discoloration, tattoos, freckles, birthmarks, moles or other skin abnormality, that may impair assessment of skin as judged by the clinician
2. Known allergic reactions to components of the Prevena Dressing, DeRoyal Incisional dressing, Hibiclens or a history of skin irritation allergic reaction to chlorohexidine, isopropyl alcohol, chlorohexidine gluconate, or silver.
3. History of skin irritation, skin sensitivity or skin disease including psoriasis, eczema, atopic dermatitis, and skin cancer.
4. Pregnant or lactating female

Lifestyle Limitations during the Study:

During this study, participants are asked to adhere to following lifestyle limitations:

* Abstain from strenuous exercise activity such as running, playing contact sports, biking, and yard work. Participants may walk at a slow pace.
* To keep both dressings shielded from sunlight and fluorescent light (e.g. wear pants or cover with elastic bandage)
* To protect dressing and not expose to high moisture/water submersion environment.
* Limit showering to once per day
* To keep the NPWT devices on and connected to dressing at all times except when showering and changing clothes

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2024-02-26 (Actual); Primary Completion 2024-03-07 (Actual); Study Completion 2024-03-07 (Actual)

PRIMARY OUTCOMES:
Change in Skin Irritation Score | Day 1 (Baseline) and Day 7
  Skin assessment is performed utilizing the Federal Drug Administration's Combined Evaluation of Skin Irritation and Sensitization utilized by the FDA for assessing topical delivery systems (https://www.fda.gov/media/117569/download). The assessments include photographs of the skin to document any noticeable differences between the two interventions visually.
  The dermal response score has eight levels between 0 and 7: 0:No evidence of irritation and 7: Strong reaction spreading beyond the dressing. Refer to the linked document for the entire scale
  The Other Effects Score (if present) has six characteristics associated with a numerical value: A(0): Slightly glazed appearance, B(1): Markedly glazed appearance, C(2): Glazing with peeling & cracking, F(3): Glazing with fissures, G(3): Film of dried serous exudates covering all or part of the dressing site, H(3): Small petechial erosions and scabs.
  The sum of the two scores represents the total irritation score.

SECONDARY OUTCOMES:
Change in skin flora bioburden | Performed Day 1 (Baseline) and Day 7
  Sterile skin swabs will be performed on approximately a 1 by 1 inch area of the knee cap on day 1 after skin prep and day 7 after removal of the dressings. Swabs will undergo bioburden testing to recover any organisms present on the skin. Day 0 assessments confirms the efficacy of the skin preparation procedure and day 7 measurements reflect rebound of skin flora under the two interventions.
Dressing Discomfort Assessment | Assessment performed once a day for 7 days by participant
  Healthy volunteer self assessment using a visual analogue scale to rate pain/discomfort experienced during study. Volunteers will mark on a 10 cm line their assessment of discomfort. No pain or discomfort indicated by a score of 0. Extreme pain or discomfort indicated by a score of 10.
Intervention Tolerance Assessment | Assessment performed once a day for 7 days by participant
  Healthy volunteer self assessment using a visual analogue scale to rate tolerance of each intervention during the study. Tolerance includes assessment of sound and impact on daily life. Volunteers will mark on a 10 cm line their assessment of discomfort. A score of 0 indicates intervention completely tolerable, does not interfere with daily living. A score of 10 indicates intervention completely intolerable, makes daily living impossible.
Change in Dressing Lift Incidence (Participant Assessment) | Assessment performed once a day by participant for Days 1 - 6. Clinician performs assessment at Day 7
  Calculate incidence rate of any dressing lift (lift or rolling) that occurs with each dressing
Change in Dressing Lift Incidence (Clinician Assessment) | Clinician performs assessment at Day 7
  Calculate incidence rate of any dressing lift (lift or rolling) that occurs with each dressing
Change in Dressing Lift Percentage (Participant Assessment) | Assessment performed once a day by participant for Days 1 - 6.
  The participant or clinician research uses a dressing diagram to indicate dressing lift or damage. Final analysis will calculate the percent area where damage occurred. A separate photograph of the dressing will confirm final assessment.
Change in Dressing Lift Percentage (Clinician Assessment) | Clinician performs assessment at Day 7
  The participant or clinician research uses a dressing diagram to indicate dressing lift or damage. Final analysis will calculate the percent area where damage occurred. A separate photograph of the dressing will confirm final assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Principal Investigator, Principal Investigator — Lincoln Memorial University
Locations (1):
- Lincoln Memorial University; Cedar Bluff Campus, Knoxville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Guidance Document defining Skin irritation and sensitization scale used as primary outcome — https://www.fda.gov/media/117569/download